CLINICAL TRIAL: NCT01979458
Title: Pilot Study to Evaluate Photometric Stereo Endoscopy (PSE) as a Tool for Imaging the Rectum and Colon
Brief Title: Photometric Stereo Endoscopy (PSE) as a Tool for Imaging the Rectum and Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Norman Nishioka, MD, Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013P001115
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2014-09

CONDITIONS: Colonic Polyps
Keywords: Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSE (Experimental): Patients whose distal colon is imaged using the PSE device. This is a pilot trial of 30 patients.
  Interventions: Device: PSE

INTERVENTIONS:
Device: PSE
  Other Names: photometric stereo endoscopy

SUMMARY:
The goal of this research is to assess photometric stereo endoscopy (PSE) as an endoscopic imaging technique. Specifically, topographical surface contrast reconstructed from the PSE data will be compared to conventional imaging contrast to assess if PSE provides enhanced contrast of abnormal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a routine colonoscopy screening
* Patients must be over the age of 18
* Patients must be able to give informed consent

Exclusion Criteria:

* Patients with bleeding/hemostasis disorders
* Patients that are pregnant
* Patients taking any anti-coagulants that would preclude them from undergoing a standard of care colonoscopy, such as Coumadin and Plavix, at the time of the study
* Patients with known colitis or active bleeding will be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Image Contrast | Immediate
  Comparison of image contrast obtained using standard colonoscopy and PSE.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States